CLINICAL TRIAL: NCT04039737
Title: Clinical Study of Qingpeng Ointment in Treating Shoulder Syndrome During Rehabilitation Period of Cerebral Hemorrhage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JDZX2015224
Record Dates: First submitted 2019-07-23; First posted 2019-07-31 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: The Efficacy of Qingpeng Ointment
Keywords: Qingpeng Ointment; Shoulder Syndrome; Rehabilitation Period of Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Take Qingpeng ointment (produced by Tibet Qizheng Tibetan Medicine Co., Ltd.) and apply it evenly on the shoulder joints, wrist joints and palms of the upper limbs. Press for 20 minutes and have rehabilitation training afer 10 minutes.
  Interventions: Drug: Qingpeng Ointment
- Control Group (No Intervention)

INTERVENTIONS:
Drug: Qingpeng Ointment — Take Qingpeng ointment (produced by Tibet Qizheng Tibetan Medicine Co., Ltd.) and apply it evenly on the shoulder joints, wrist joints and palms of the upper limbs. Press for 20 minutes and have rehabilitation training afer 10 minutes.
  Arms: Treatment Group

SUMMARY:
A randomized, controlled study is conducted. 120 patients with post-stroke shoulder-shoulder syndrome who meet the inclusion criteria are randomized into treatment group and control group, 60 patients in each group. The treatment group is treated with Qingpeng ointment. The goal of this trial is to verify the clinical efficacy of Tibetan medicine Qingpeng ointment in improving post-stroke shoulder-hand syndrome, and to investigate its effect on pain level, swelling degree, hand movement function, activity and activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for stroke;
2. Meet the diagnostic criteria for shoulder-hand syndrome, stage I
3. The course of disease is between 15 days and 6 months;
4. Consciousness, no serious cognitive impairment, with examination and treatment;
5. Age between 20 and 80 years old;
6. Sign the informed consent form and volunteer to participate in the study.

Exclusion Criteria:

1. Repeated stroke patients or shoulder-hand syndrome patients with repeated attacks or exacerbations;
2. The course of stroke is >6 months;
3. Those with serious heart, liver and kidney diseases and moderate to severe infections;
4. Unconsciousness or a combination of incompetent cognitive impairment and complete aphasia.
5. Take painkillers or other treatments that treat shoulder pain.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Painful degree change of ipsilateral shoulder | VAS will be tested before treatment and after a 4-week treatment so as to compare the efficacy.Twice in total
  Visual analog scale(VAS) is used to test the painful degree. It contains 0-10 scores,while "0"means no pain, "10"means most severe painful.The higher the scores,the more painful.
Motor function change | This scale will be tested before treatment and after a 4-week treatment so as to compare the efficacy.Twice in total
  Using Simplified Fugl-Meyer motion function assessment method to assess the motor function of affected side.The total score of Fugl-Meyer motor function assessment scale is 100 points，50 items intotal with 2 points each. Accordding to the quality of mission completion，evaluater mark score of "0","1",2".Among them, 33 items are evaluated for upper limbs, with a total score of 66 points. And 17 items are evaluated for lower limbs,with a total score of 34 points.The higher the scores, the better motor function.If the total score is less than 50, it means severe dyskinesia.If the total score is between 50-84, it means obvious movement disorder.If the total score is between 85-95, it means moderate dyskinesia.If the total score is between 96-100, it means mild dyskinesia.
Activity of daily living change (ADL) | This scale will be tested before treatment and after a 4-week treatment so as to compare the efficacy.Twice in total
  Using Modified Barthel Index to assess the activity of daily living. TheMBI scale includes 11 items with total scores of 100. Evaluation is based on the actual situation of the patient.The sum of the scores of each item is the total score,and the lowest score is"0",the highest scores is"100".If the scores is between 0-20 points,it means extremely severe dysfunction.If the scores is between 25-45 points,it means severe dysfunction.If the scores is between 50-70 points it means moderate functional defects.If the scores is between 75-95 points,it means mild functional defects.If the scores is 100 points,it means ADL self-care.The higher the total scores,the better the ADL.
Shoulder joint mobility change | These will be tested before treatment and after a 4-week treatment so as to compare the efficacy.Twice in total
  Test the shoulder joint mobility with a protractor.The movements of the shoulder joints are as follows:Flexion：70-90°；Stretch：40°；Outreach：80-90°；Adduction：40-60°；Pronation：70-90°；External rotation：15°；Lift up：160-180°.The bigger the degrees，the better the shoulder joint mobility.

SECONDARY OUTCOMES:
Safety evaluation | After 4 weeks of treatment, evaluate adverse reactions and make a record.
  Safety rating includes 4 levels.Level 1 means "Safe, without any adverse reactions".Level 2 means "Safer, if there is an adverse reaction, you can continue treatment without any treatment ".Level 3 means " Have safety problems, have moderate adverse reactions, and continue treatment after treatment". Level 4 means " Suspension test due to adverse reactions".

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Chen, Master, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese medicine, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Pan R, Ling S, Yang H, Huang Y, Zhan L, Zhong Y, Chen H. Clinical Study of Qingpeng Ointment Treating Shoulder-hand Syndrome After Cerebral Hemorrhage During the Rehabilitation Period. Comb Chem High Throughput Screen. 2021;24(7):968-975. doi: 10.2174/1386207323666201211093227. PMID 33308122